CLINICAL TRIAL: NCT01622907
Title: European Multicenter Study Using Hybrid Staged Operating Room and Interventional Catheter Ablation Techniques to Treat Chronic AF
Brief Title: Hybrid Staged Operating Room and Interventional Catheter Ablation for Atrial Fibrillation
Acronym: HISTORIC-AF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Collaborators: Meditrial SrL (Industry)
Responsible Party: Principal Investigator, Claudio Muneretto, M.D., Professor. Director, Department of Cardiac Surgery, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Other Study IDs: HISTORIC AF 2011-10-11
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Atrial Fibrillation
Keywords: Catheter ablation, radiofrequency; Epicardially applied radiofrequency ablation; Minimally invasive surgical approach
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pts Symptomatic Recurrent Persistent AF: Patients with Symptomatic Recurrent Persistent AF or Long standing AF,for > 1-year < 5 years duration

SUMMARY:
Prospective, multi-center, investigator-driven trial. This study hypothesizes that combining surgical endoscopic and transcatheter techniques in a staged fashion provides superior clinical outcomes than isolated surgical/EP approaches in patients with persistent AF lasting > 1 year but > 5 years.

The proposed procedure involves the creation of cardiac lesions with epicardially applied radiofrequency (RF) ablation through a minimally invasive surgical (MIS) approach followed by a delayed EP ablation procedure performed at 1-2 months from the surgical operation.

DETAILED DESCRIPTION:
New ablative technologies have been developed to simplify the original "cut and sew" Cox Maze procedure so that it can now be used for routine treatment of AF in patients undergoing open-heart surgery, as well as in a stand-alone arrhythmia procedure. A minimally invasive, thoracoscopic surgical treatment of AF is able to address both the triggers for AF by pulmonary vein isolation and the left posterior atrial wall exclusion, which after the pulmonary veins is the next most important atrial substrate in the promotion of AF.

New hybrid procedures attempt to combine the success rate and the minimally invasive nature of thoracoscopic mini-Maze with the effectiveness and short recovery times associated with catheter ablation. The key is blocking signals that cause the arrhythmia from both outside (epicardial) and inside (endocardial) the heart.

Suboptimal results of both catheter ablation and surgery suggest that success in the treatment of long standing persistent AF and persistent lone AF will benefit from a close collaboration between the cardiothoracic surgeon and the electrophysiologist, to offer patients the best available combination of treatments for any given set of cardiovascular lesions.

Hybrid treatment for AF is being increasingly adopted in Europe and the United States and has been assessed for the treatment of AF at the Coordinating Center (Brescia, Italy) with promising results.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be treated initially by thorocoscopic epicardial surgical RF ablation to create a box lesion around the pulmonary veins, ganglionated plexi, and superior vena cava-inferior vena cava (SVC-IVC) connecting lesions.

Four to maximum 8 weeks following the surgical ablation procedure, the patient is returning to the EP Laboratory to:

Assess integrity of the Box lesion Eliminate gaps in the surgical lesions when found Terminate fragmented potentials Perform a Caval-Tricuspid Isthmus (CTI) lesion line Upon completion of this procedure, integrity of the lesions is reassessed just prior to withdrawing the EP catheters from the LA.

Exclusion Criteria:

* History of Recurrent Persistent or Long Standing Persistent AF for more than 5 years; Documented left atrial size (AP diameter) greater than 55 mm; Documented left ventricular ejection fraction (LVEF) of 40% or less; History of cerebrovascular disease, including stroke or transient ischemic attack (TIA) within 6 months prior to enrollment; Significant underlying structural heart disease requiring surgical or procedural intervention; Previous heart surgery; Chronic obstructive pulmonary disease (< 70% predictive lung function); Contraindication to anticoagulant therapy, or inability to comply with anticoagulant therapy; Other clinical conditions precluding inclusion (e.g., organ disease, disturbances of hemostasis, etc.); Pregnancy, planned pregnancy or breastfeeding; Concomitant cardiac surgery procedure planned.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Symptomatic Recurrent Persistent AF or Long Standing Persistent AF, defined as persistent AF for greater than 1-year but less than 5 years duration (according to the HRS/EHRA/ECAS Expert Consensus Statement on Catheter and Surgical Ablation of Atrial Fibrillation)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
PRIMARY EFFICACY ENDPOINT: 24-hour Holter monitoring | 9 months following the end of the blanking period
  The primary efficacy endpoint is the rate of therapeutic success, with a target rate of > 60%. Therapeutic success is defined as freedom from AF, during the 9 months following the end of the blanking period, based on 24-hour Holter monitor results, and freedom from AADs beginning at 6 months following surgery. The blanking period is 3 months following the surgical ablation procedure.

SECONDARY OUTCOMES:
SECONDARY EFFICACY ENDPOINTS: 24-hour Holter monitoring | 9 months following the end of the blanking period
  Rate of therapeutic success is defined as freedom from AF, 9 months following the end of the blanking period, based on 24-hour Holter monitoring. The target success rate is >60%. Rate of therapeutic success is defined as freedom from AF, during the 9 months following the end of the blanking period.The blanking period is 3 months following the surgical ablation procedure.

CONTACTS AND LOCATIONS:
Overall Officials: CLAUDIO MUNERETTO, PROF., Study Chair — UNIV. HOSP. SPEDALI CIVILI
Locations (10):
- Louis Pradel Hospital, Lyon, France
- Germany (3):
  - Heart Center Brandenburg- Immanuel, Bernau
  - Stadtische Kliniken, Dortmund
  - Hamburg Uke, Hamburg
- Italy (3):
  - Ospedale Gavazzeni, Bergamo
  - Univ. Hosp. Spedali Civili, Brescia
  - Univ.Hosp. Molinette, Torino
- University Hospital, Krakow, Poland
- United Kingdom (2):
  - Hammersmith Hospital, London
  - Royal Brompton, London

REFERENCES:
- [Background] Bisleri G, Curnis A, Bottio T, Mascioli G, Muneretto C. The need of a hybrid approach for the treatment of atrial fibrillation. Heart Surg Forum. 2005;8(5):E326-30. doi: 10.1532/HSF98.20051125. PMID 16099734
- [Derived] Muneretto C, Bisleri G, Rosati F, Krakor R, Giroletti L, Di Bacco L, Repossini A, Moltrasio M, Curnis A, Tondo C, Polvani G. European prospective multicentre study of hybrid thoracoscopic and transcatheter ablation of persistent atrial fibrillation: the HISTORIC-AF trial. Eur J Cardiothorac Surg. 2017 Oct 1;52(4):740-745. doi: 10.1093/ejcts/ezx162. PMID 29156015